CLINICAL TRIAL: NCT03623594
Title: Abdominal Trunk Function After Surgical Repair of Abdominal Rectus Muscle Diastasis: Outcome Measured With the Abdominal Trunk Function Protocol
Brief Title: Abdominal Trunk Function After Surgical Repair of Abdominal Rectus Muscle Diastasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Stockholm South General Hospital (Other)
Responsible Party: Principal Investigator, Gabriel Sandblom, Associate Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARD
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Rectus Abdominus; Diastasis, Complicating Delivery

STUDY DESIGN:
Intervention Model Description: Repair of the abdominal rectus diastasis with a double row plication using absorbable Quill
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical repair of the diastasis (Experimental): Repair of the diastasis with a double row plication using absorbable Quill suture
  Interventions: Procedure: Surgical repair of the diastasis

INTERVENTIONS:
Procedure: Surgical repair of the diastasis — Repair of the diastasis with a double row plication using absorbable Quill suture

SUMMARY:
There is insufficient evidence regarding the benefit from surgical reconstruction of post-partum abdominal rectus muscle diastasis. The purpose of this study is to evaluate the abdominal trunk function preoperatively and postoperatively in a group of women undergoing surgery for abdominal rectus muscle diastasis.

DETAILED DESCRIPTION:
There is little evidence regarding the various treatment options of abdominal rectus muscle diastasis in post-partum women. The lack of evidence may, to a great extent, be explained by the lack of uniform criteria for assessing the trunk function and how the trunk function affects the ability to perform daily activities. To be able to evaluate the condition with symptomatic ARD a more comprehensive, multimodal instrument is therefore needed.

In collaboration with the surgical clinic and the physiotherapy clinic at Södersjukhuset a multimodal examination test was developed with the purpose to be able to evaluate the full picture of the condition.

The purpose of this study was to evaluate the effect of surgical reconstruction of post-partum abdominal rectus muscle diastasis in women with insufficient improvement after adequate physical training using a novel multimodal evaluation tool.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking women
* BMI <35
* Inter-recti distance >3cm
* Lack of response to standardized core stabilizing training
* >1 year since last partus
* No intention of further pregnancies

Exclusion Criteria:

* Inability to quit smoking
* BMI >35
* Inter-recti distance <3cm
* <1 year since last partus
* Further pregnancies not excluded

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Abdominal Trunk Function assessed with Disability Rating Index (DRI) | One year
  DRI is a self -report form that covers twelve activities related to daily activities. Each activity is rated on a visual analogue scale from 0 to 100. The total score thus ranges from 0 to 1200, with higher scores corresponding to better function.

SECONDARY OUTCOMES:
Health-related quality of life: SF-36 | One year
  SF-36 is a set of generic and coherent quality-of-life measures. The form includes 36 items covering various aspects of quality of life. It gives eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The higher the score the less disability.
Urogenital distress rated with Urinary Distress Inventory Short Form (UDI-6) | One year
  The UDI-6 is a six item symptom inventory, specific to symptoms associated with lower urinary tract dysfunction, and combines information on irritative, stress and obstructive symptoms. It was developed for self-administration and is intended to be used in combination with IIQ-7. Patients rate how much they experience impaired function of urinary incontinence and the extent to which urinary incontinence affects daily functioning with four response options per item. The mean score of items is multiplied by 33 1/3 to convert to a 0-100 scale. Higher scores indicate more symptom distress.
Urinary stress incontinence rated with IIQ-7. | One year
  The IIQ-7 is a seven item life-impact assessment instrument specific to UI, and covers separate domains of physical activity, travel, social, and emotional health. It was developed for self-administration and is intended to be used in combination with UDI-6. Patients rate how much they experience impaired function of urinary incontinence and the extent to which urinary incontinence affects daily functioning with four response options per item. The mean score of items is multiplied by 33 1/3 to convert to a 0-100 scale. Higher scores indicate more impact on daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Sandblom, Ass Prof, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No